CLINICAL TRIAL: NCT03899948
Title: Teacher Anxiety Program for Elementary Students
Acronym: TAPES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Responsible Party: Principal Investigator, Golda S. Ginsburg, Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 18-004-6; R324A170071 (Other Grant/Funding Number: Institute of Education Sciences)
Record Dates: First submitted 2019-03-28; First posted 2019-04-02 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Anxiety
Keywords: Excessive Anxiety; Teacher Training; Elementary School; School-based; Effectiveness Research; Randomized Controlled Trial
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This study uses a parallel Randomized Controlled Trial Design. Following teacher enrollment, randomization occurs at the teacher level with a 1:1 (20 TAPES condition: 20 TAT condition) ratio. Teachers in each condition complete the training and intervention concurrently.
Who Masked: Outcomes Assessor
Masking Description: Independent Evaluators (IEs) conduct all post and follow-up assessments. These IEs are blind to the condition of all participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teacher Anxiety Program for Elementary Students (TAPES) (Experimental): Teachers in the experimental condition attend a 6-hour training on the TAPES program. The teachers learn to implement a brief intervention (5 meetings) with the student and his or her parent, utilize classroom anxiety-reduction strategies, and apply relationship enhancement strategies to improve the relationship with the target student and parents.
  Interventions: Behavioral: Teacher Anxiety Program for Elementary Students
- Teacher Anxiety Training (TAT) (Active Comparator): Teachers in this condition receive training about childhood anxiety and classroom anxiety-reduction strategies using a 3-hour typical teacher professional development training format.
  Interventions: Behavioral: Teacher Anxiety Training

INTERVENTIONS:
Behavioral: Teacher Anxiety Program for Elementary Students — TAPES consists of three core components: 1) training in evidenced-based anxiety reduction strategies that teachers will implement to identify and assist specific anxious students and classroom-wide strategies helpful to all students, 2) evidenced-based material for teachers to review with parents regarding how to reduce student anxiety at home, thus improving school-home communication and shared goals and 3) training in how to conduct 5 brief (30 minute) teacher-parent-student meetings to teach and practice the TAPES anxiety-reduction strategies.
  Other Names: TAPES
  Arms: Teacher Anxiety Program for Elementary Students (TAPES)
Behavioral: Teacher Anxiety Training — The TAT is a 3-hour professional development training for teachers. Training focuses on recognizing the signs and symptoms related to child anxiety and utilizing classroom-wide strategies to help reduce anxiety in the classroom.
  Other Names: TAT
  Arms: Teacher Anxiety Training (TAT)

SUMMARY:
The purpose of the study is to compare two teacher trainings developed to assist elementary students who struggle with excessive anxiety. The goal of both teacher trainings is to improve teachers' knowledge and skills for identifying and assisting students with excessive anxiety. The first training program is called TAPES (Teacher Anxiety Program for Elementary Students) and involves a 6 hour teacher training. Teachers in this training program will implement anxiety reduction skills in the classroom and complete 5 brief (approximately 30 minute) meetings with the student and his or her parent(s)/guardian(s). The second training program, Teacher Anxiety Training (TAT), involves a 3 hour teacher training. Teachers in the TAT condition learn to implement anxiety reduction skills in the classroom, but do not conduct individual meetings with parents and students. The investigators do not know if TAT and TAPES work equally well, or if one is better than the other. Both will be administered by teachers to see if they help youth with excessive anxiety feel less worried.

DETAILED DESCRIPTION:
Summary, Benefit to Stakeholders, and Aims: Teachers lack the knowledge and skills to support the learning of students with excessive anxiety who have, or at risk of developing, an identified disability. Excessive student anxiety is a common problem that severely impairs short and long term academic functioning and increases teacher burden. Conversely, reducing student anxiety has been associated with improvement in educational functioning. Because anxiety manifests daily in the classroom, teachers are in an ideal position to identify and help students manage their anxiety. One universal intervention for anxiety reduction exists, but its feasibility and efficacy are not established. The aims of this project are to address this gap in teacher training. Specifically, the aims of this proposal include: Aim 1) to develop the Teacher Anxiety Program for Elementary Students (TAPES) and assess its usability, acceptability and feasibility; Aim 2) to determine whether teachers can implement TAPES with high fidelity and quality; Aim 3) to examine the impact of TAPES, compared to a standard professional development condition, on teacher a) knowledge and b) use of anxiety reduction strategies with students with excessive anxiety (Primary Outcomes); and Aim 4) to examine the impact of TAPES on student outcomes. Exploratory aims will examine the mediators, predictors, and moderators of TAPES impact on teachers' knowledge and skill. If effective, TAPES has the potential to directly benefit: 1) teachers--by providing training in an important and relevant, but neglected area that will enhance their professional development and effectiveness in the classroom; and 2) children--by reducing their anxiety and improving their educational, social, and behavioral functioning.

Description of TAPES: The proposed teacher training is appropriate for elementary teachers to enhance their capacity to support students with excessive anxiety. The training includes one full day of instruction, materials to use with individual students and their parents (in 5 meetings), and guidelines for classroom-wide strategies to reduce anxiety. The section below describes 1) the content of the teacher training and supportive empirical evidence, 2) how this training differs from current teacher practices for anxious students, 3) a proposed theory of teacher and child behavior change and 4) evidence supporting the feasibility of implementing TAPES in an authentic school environment. This teacher training is not intended to replace or change the role of existing mental health providers or other members of schools' interdisciplinary teams. Given that teachers are members of an interdisciplinary team, the study team will obtain input from school personnel to ensure that the teacher-training fits within the goals/mission of the interdisciplinary team.

Description of TAPES content: Overview: The primary goal of TAPES is to enhance teachers' capacity to identify and reduce anxiety in their students. Toward this end, the proposed content of TAPES consists of three core components: 1) training in evidenced-based anxiety reduction strategies that teachers will implement to identify and assist specific anxious students and classroom-wide strategies helpful to all students, 2) evidenced-based material for teachers to review with parents regarding how to reduce student anxiety at home, thus improving school-home communication and shared goals and 3) training in how to conduct conjoint teacher-parent-student meetings to improve the quality of the teacher-parent-student relationship. Each component is described below.

Training and Evidence Related to Child Anxiety Reduction Skills: Teachers will learn skills based on cognitive behavioral strategies (CBT) including relaxation training (to reduce physiological arousal), behavioral strategies (e.g., "exposure" or facing anxiety provoking situations which lowers anxiety via new learning), addressing maladaptive thoughts that maintain anxiety, and problem solving skills. To implement these new skills with specific children teachers will be trained to use a school-home journal that includes a type of daily report card that tracks behavioral exposures and use a reward system for increasing brave behavior /adaptive coping skills.). These "common elements" of CBT are powerful agents of change and have been implemented by CBT experts and non-experts. As such, these skills are established and empirically-supported; however, they have not been evaluated when delivered by teachers.

Teachers will also receive training in effective classroom-based accommodations that may be needed (e.g. untimed testing) or may need to be gradually faded if they are maintaining anxiety through negative reinforcement (e.g. allowing child to avoid participating in class due to anxiety). Another component of the teacher training includes skills that teachers deliver to their classroom (i.e., such as leading the entire class in a relaxation exercise prior to an exam; teacher using a coping model or teacher reducing their accommodation of avoidant/anxious behavior for all students). Finally, teachers will be trained in how to modify their own behaviors that have been shown to increase student anxiety (e.g., hostility, over-control). These modifications are also designed to improve the quality of the teacher-student relationship. Research on the role of teacher behavior in the development and/or maintenance of child anxiety suggests that teachers who exhibit highly controlling behaviors, such as issuing frequent directives, tend to increase child anxiety and negatively affect children's ability to learn. Conversely, positive teacher-child relationships have been found to protect youth from developing internalizing behavior problems over time. Consequently, TAPES aims to modify these teacher behaviors.

Training and Evidence Related to Conjoint Parent-Teacher-Student Meetings. Training teachers in conducting conjoint meetings will enhance teachers' ability to formalize mechanisms for sharing information about anxiety reduction and will enhance communication and relationship quality between parent, teacher, and student. Training in these conjoint meeting will also allow the teacher to clarify roles and responsibilities with respect to helping the child, and devise a collaborative plan with similar language and tools to facilitate generalization of skills between school and home. Implementation of this component will involve approximately 5 conjoint-30 minute meetings over an 8 week period. During these meetings, parents, students, and teachers will create and modify anxiety hierarchies, mutually decide on practice tasks, and develop a contingency management plan. Target behaviors are individualized based on the needs of the child (e.g., raising a hand to answer a question in class for a child with social anxiety; separating from parents for a child with separation anxiety). These meetings can be supplemented by phone and email contacts between teacher and parents/students as needed.

TAPES Training Format and Implementation: Students' primary teacher will participate in a one-day training (approximately 6 hours). One of the most important strategies for ensuring that TAPES is implemented with high fidelity is appropriate training and ongoing consultation. Training strategies will be based on published guidelines and will include active/experiential learning strategies, opportunities for observation (via video clips), live modeling and role plays, and coached practice. Ongoing performance feedback and consultation has been found to enhance learning and is related to higher fidelity. Thus, teachers will be offered 30-minutes of weekly consultation by the PIs for each active TAPES students. Consultation will include case review, skill rehearsal, problem-solving obstacles, and feedback regarding performance based on audiotaped sessions. Meetings will be held in person, over the phone, or via Skype at times convenient for teachers. After each teacher identifies their first child, the PIs will attend one conjoint meeting in order to provide performance feedback (all conjoint meetings are audiotaped for fidelity). The PIs will also provide in classroom coaching for 30-minutes for each student enrolled. Training materials will be available on the internet or thumb drive for reference.

Research Plan Overview: Design and Methods. This three-year development project consists of 3 stages. Stage one (months 1-6) involves establishing a Development Team (DT) that will review the initial draft of TAPES and provide feedback to ensure that TAPES is acceptable to teachers and feasible for the school setting. Stage two (months 7-20) involves two successive open trials of the TAPES protocol with 15 teachers and 20 children. This stage will allow for "trial runs" of the training to assess feasibility, acceptability and utility of the training. Data and qualitative feedback gleaned during the first open trial will inform modifications for the second open trial. The investigators will present and discuss data with the DT after each open trial. Study staff will also ask 5 teachers from open trial 1 to test out the revisions for open trial 2. Based on knowledge gained in this stage, appropriate modifications will be made for stage three. Stage three (months 21-34) involves a pilot Randomized Controlled Trial (RCT) using a randomized controlled design comparing TAPES to the Teacher Anxiety Training (TAT). TAT (developed by the PIs for use in other studies and described below) will be used to represent "typical" teacher professional development training. The RCT will be conducted in three phases. Phase 1 consists of recruiting, randomizing, and training teachers in either TAPES or TAT. Also during this phase (but after the training), teachers will recruit anxious children and study staff will screen and evaluate them to determine eligibility. In Phase 2 teachers will implement TAPES or TAT. Phase 3 involves a post-intervention (after 8 weeks) and a three-month follow-up assessment of the primary (teacher behavior) and secondary (child) outcomes. Trained independent evaluators (IEs) will assess primary outcomes (teacher behavior). The culmination of these iterative stages will be a final version of the training that will be ready for evaluation in a larger efficacy trial.

Detailed Description of Each Stage Stage 1: Establish DT and refine initial version of the TAPES Protocol. The DT will strive to ensure that the teacher training will be acceptable, feasible, and usable in the school setting. The DT will consist of the PIs, two national experts in teacher training, two experts in school-home collaborative interventions, and two experts in training school-based personnel in CBT techniques for anxious youth. A CT school psychologist and two CT elementary teachers will complete the DT. DT members will provide detailed feedback about the TAPES strategies, study methods/measures, perceived barriers to successful implementation and adoption by teachers, and solutions to potential barriers. Information from this meeting will be used to revise the protocol in preparation for the first open trial as well as successive phases of the study.

Stage 2: Open Trials. During Stage 2, teachers and IEs will be trained, and the study team will conduct two sequential open trials. Study staff will engage in screening activities of students and IEs will complete baseline evaluations on referred students. The purpose of the open trials is to evaluate the feasibility of the training, modify methods as needed, allow teachers to implement the skills learned in the training and receive real time coaching and consultation with anxious children. Data on TAPES usability, acceptability, fidelity, satisfaction, and teacher and child outcomes will also be collected. After each open trial, feedback (via exit interviews and standardized measures) from teachers, students, and parents will be integrated by the research team and presented to the DT for another revision of the protocol. Teachers will be asked to participate in an exit interview after they implement TAPES with an anxious child.

Stage 3: Pilot RCT. In stage 3, the study team will conduct a pilot RCT with 40 teachers and a maximum of 60 anxious youth. The RCT will be conducted in 3 phases.

Phase 1 - Recruitment, Randomization, Training, Student Screening, and Baseline Evaluations: In Phase 1, teachers will be randomly selected from the pool of interested participants and randomized to TAPES or TAT. Once randomized, teachers will complete their assigned training. Teachers will then identify potentially eligible students from their classes and provide information about the study to their parents. Interested parents will contact study staff and complete a brief phone screen. Students who appear eligible based on the phone screen (e.g., have elevated anxiety; are in elementary school) will be invited to complete informed consent and a full baseline evaluation with an IE. Families who meet criteria on the baseline evaluation will be considered eligible (see Inclusion/Exclusion criteria).

Phase 2 - TAPES/TAT Implementation: Teachers will implement TAPES or TAT depending on their random assignment over 8 weeks from child enrollment.

Phase 3 - Post- and Follow-up Evaluations: At the end of the 8 weeks, teachers and children in both groups will complete a post evaluation. Teachers, students, and parents will complete a TAPES satisfaction measure and provide feedback to enhance the protocol. Teachers will complete an exit interview. Students who need mental health services will be referred to the school counselor or community provider for treatment. A 3 month follow-up evaluation to assess sustained use of TAPES/TAT skills will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Must attend a CT elementary school
* Must have elevated anxiety symptoms, which is defined as a total Spence Children's Anxiety Scale t score > 60 based on parent and/or child report and/or a Clinician Severity Rating (CSR) of 3 or greater on the Anxiety Disorder Interview Schedule (ADIS-V).

Exclusion Criteria:

* Any medical or psychiatric condition contraindicating the study participation (based on clinical interview; such as recent suicidality)

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline on the Teacher Knowledge Assessment | Baseline, 8 week Post-Intervention
  Two equivalent forms assessing teachers' knowledge of anxiety symptoms and anxiety-reduction strategies. Comprised of multiple-choice and short-answer questions.
Change from Baseline on the Classroom Observation of Teachers Skills | Baseline, 8-week post-intervention, 3-month post-intervention follow-up
  This is a form created for this study that is completed by two independent evaluators following direct observations of teachers. Observers rate the teachers' use of teaching behaviors reviewed in the training. Scores are generated for 3 domains: Teacher behaviors that may decrease anxiety (Do Behaviors), behaviors that may increase anxiety (Don't Behaviors), and behaviors that evidence strong teacher-student relationships (Relationship Behaviors). Teachers are rated on a 5 point Likert-type scale, with 0 indicating poor behavior and 4 indicating very good or excellent behavior (min score = 0, max score = 4 on all domains). There is no combined total score. Higher values in each domain demonstrate greater mastery of teaching behaviors reviewed in the training.

SECONDARY OUTCOMES:
Change from Baseline on the Modified Anxiety Diagnostic Interview Schedule, for the Diagnostic and Statistical Manual Fifth Edition (ADIS-V) | Baseline, 8-week post-intervention, 3-month post-intervention follow-up
  Semi-structured clinical interview assessing student anxiety diagnosis and severity.
Change from Baseline on the Spence Children's Anxiety Scale, Child and Parent Versions | Baseline, 8-week post-intervention, 3-month post-intervention follow-up
  The Spence Children's Anxiety Scale is a reliable and valid measure of anxiety symptoms in children. Both versions use a 4-point Likert scale to assess frequency of symptoms (0 = never, 3 = always). The child report has 44 items--38 of which are used to calculate the total score. The parent report has a total of 39 items--38 of which are used in the total score (minimum score 0 , maximum score 114). On both forms, higher scores represent higher levels of anxiety.
Change from Baseline on the Child Anxiety Impact Scale, Child and Parent Versions (& adapted Teacher Version) | Baseline, 8-week post-intervention, 3-month post-intervention follow-up
  The Child Anxiety Impact Scale measures the impact of a child's anxiety across school, home, and social domains. Both versions use a 4-point Likert scale (0 = not at all, 3 = very much) to assess the frequency of anxiety impairment in various areas. The range for the total score is 0 (minimum) to 81 (maximum). Subscale scores range from a minimum of 0 to a maximum of 30, 33, and 18 for the school, social, and home subscales, respectively. Higher scores represent greater interference of anxiety in child functioning.
Change from Baseline on the Woodcock Johnson IV Tests of Achievement (Fluency subtests) | Baseline, 8-week post-intervention, 3-month post-intervention follow-up
  Psychometrically validated measure of academic fluency in children. Scores are generated as standard scores with a mean of 100 and a standard deviation of 15. Higher scores represent better academic performance.
Change from Baseline on the Woodcock Johnson IV Tests of Cognitive Abilities (Numbers Reversed subtest) | Baseline, 8-week post-intervention, 3-month post-intervention follow-up
  Psychometrically validated measure of working memory in children. Scores are generated as standard scores with a mean of 100 and a standard deviation of 15. Higher scores represent better working memory capacity.
Change from Baseline on the Family Accommodation Scale, Anxiety (FASA) Parent form (& adapted teacher version) | Baseline, 8-week post-intervention, 3-month post-intervention follow-up
  Measures frequency of parent (and teacher) accommodation behaviors in relation to child's anxiety symptoms. Items are rated on a 5-point Likert scale (0 = Never, 4 = Daily). Items 1-9 are summed to find total accommodation behaviors (minimum score = 0, maximum score = 36). Higher scores represent more accommodation behaviors associated with more anxiety-related impairment in family functioning or classroom functioning.
Change from Baseline on the Children's Global Assessment Scale (CGAS) | Baseline, 8-week post-intervention, 3-month post-intervention follow-up
  The Children's Global Assessment Scale is a single-item measure of child's overall behavioral functioning assigned by a clinical interviewer. Scores on this scale range from 1 to 100. Higher scores are associated with more adaptive functioning. More specifically, scores below 70 are indicative of increasingly severe impairment in behavioral functioning.
Change from Baseline on the Clinical Global Impression - Severity (CGI-S) and Improvement (CGI-I) Scales | Baseline, 8-week post-intervention, 3-month post-intervention follow-up
  These two single-item scales measure a student's anxiety symptom severity and improvement as rated by a clinical interviewer. On the Severity scale, scores range from 1 (Normal) to 7 (Extremely Ill). Higher scores represent greater anxiety symptom severity. On the Improvement scale, scores range from 1 (Very Much Improved) to 7 (Very Much Worse). Lower scores represent better outcomes relative to the baseline assessment.
Change from Baseline on the School Anxiety Scale | Baseline, 8-week post-intervention, 3-month post-intervention follow-up
  The School Anxiety Scale is a teacher-report measure of anxiety symptoms exhibited in the classroom. This 16-item measure uses a 4-point Likert scale to measure the frequency of anxiety-related behaviors (0 = never, 3 = always). The scale has a minimum score of 0, and a maximum score of 48. Higher scores represent more frequent anxiety-related behaviors in the classroom.

CONTACTS AND LOCATIONS:
Overall Officials: Golda S Ginsburg, PhD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, West Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cartwright-Hatton S, Mather A, Illingworth V, Brocki J, Harrington R, Wells A. Development and preliminary validation of the Meta-cognitions Questionnaire-Adolescent Version. J Anxiety Disord. 2004;18(3):411-22. doi: 10.1016/S0887-6185(02)00294-3. PMID 15125986
- [Background] Drake KL, Ginsburg GS. Parenting Practices of Anxious and Non-Anxious Mothers: A Multi-method Multi-informant Approach. Child Fam Behav Ther. 2011;33(4):299-321. doi: 10.1080/07317107.2011.623101. Epub 2011 Dec 6. PMID 22639487
- [Background] James AC, James G, Cowdrey FA, Soler A, Choke A. Cognitive behavioural therapy for anxiety disorders in children and adolescents. Cochrane Database Syst Rev. 2013 Jun 3;(6):CD004690. doi: 10.1002/14651858.CD004690.pub3. PMID 23733328
- [Background] Assor A, Kaplan H, Kanat-Maymon Y, Roth G. Directly controlling teacher behaviors as predictors of poor motivation and engagement in girls and boys: The role of anger and anxiety. Learning and Instruction 15(5): 397-413, 2005.
- [Background] O'Connor EE, Dearing E, Collins BA. Teacher-child relationship and behavior problem trajectories in elementary school. American Educational Research Journal 48(1):120-62, 2011.
- [Background] Beidas RS, Kendall PC. Training Therapists in Evidence-Based Practice: A Critical Review of Studies From a Systems-Contextual Perspective. Clin Psychol (New York). 2010 Mar;17(1):1-30. doi: 10.1111/j.1468-2850.2009.01187.x. PMID 20877441
- [Background] Fixsen DL, Naoom SF, Blase KA, Friedman RM. Implementation research: A synthesis of the literature. Tampa, FL: University of South Florida, Louis de la Parte Florida Mental Health Institute, The National Implementation Research Network, 2005.
- [Background] Sholomskas DE, Syracuse-Siewert G, Rounsaville BJ, Ball SA, Nuro KF, Carroll KM. We don't train in vain: a dissemination trial of three strategies of training clinicians in cognitive-behavioral therapy. J Consult Clin Psychol. 2005 Feb;73(1):106-15. doi: 10.1037/0022-006X.73.1.106. PMID 15709837
- [Derived] Ginsburg GS, Pella JE, Piselli K, Chan G. Teacher Anxiety Program for Elementary Students (TAPES): intervention development and proposed randomized controlled trial. Trials. 2019 Dec 30;20(1):792. doi: 10.1186/s13063-019-3863-9. PMID 31888726

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-06): https://cdn.clinicaltrials.gov/large-docs/48/NCT03899948/Prot_SAP_000.pdf